CLINICAL TRIAL: NCT02736578
Title: Intraoperative Pancreatic Cancer Detection Using Multimodality Molecular Imaging
Brief Title: Cetuximab-IRDye 800CW and Intraoperative Imaging in Finding Pancreatic Cancer in Patients Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistics
Sponsor: Eben Rosenthal (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Professor of Otolaryngology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-35789; NCI-2016-00433 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PANC0024 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cetuximab IRDye800, 50 mg (Experimental): On day 0, participants receive a 100 mg cetuximab loading dose by intravenous infusion (IV), followed 1 hour later by cetuximab-IRDye 800CW IV at 50 mg, followed by surgery with intraoperative imaging within 2 to 5 days.
  Interventions: Drug: Cetuximab-IRDye800; Drug: Cetuximab
- Cetuximab IRDye800, 100 mg (Experimental): On day 0, participants receive a 100 mg cetuximab loading dose by intravenous infusion (IV), followed 1 hour later by cetuximab-IRDye 800CW IV at 100 mg, followed by surgery with intraoperative imaging within 2 to 5 days.
  Interventions: Drug: Cetuximab-IRDye800; Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab-IRDye800 — Administered intravenously (IV) at 50 or 100 mg
  Other Names: Cetuximab-IRDye 800CW
Drug: Cetuximab — Administered as a 100 mg IV loading dose
  Other Names: Erbitux; C225

SUMMARY:
This phase 1-2 trial studies the side effects and best dose of cetuximab-IRDye 800CW when used with intraoperative imaging, to determine the utility of cetuximab-IRDye 800CW to identify and assess pancreatic cancer in patients undergoing surgery to remove the tumor. Cetuximab-IRDye 800CW may help doctors better identify cancer in the operating room by making the cancer visible when viewed through a fluorescent imaging system.

DETAILED DESCRIPTION:
This is a dose-escalation study of 50 mg or 100 mg cetuximab-IRDye800.

Clearance of the tumor margin during surgical resection of pancreatic cancer is clinical importance, as margin-positive resections are suspected to be associated with rapid emergence of distant metastases shortly after surgery. However, pancreatic cancer is known to be difficult to visualize intraoperatively. Nonetheless, better detection of tumor tissue might improve the rate of complete tumor clearance, thereby improving outcomes. However, in order to be actionable, the data from such enhanced tumor detection must be available during the resection procedure. This study evaluates the use of a dye, Cetuximab-IRDye 800CW, that is administered pre-surgery, and is detectable during the surgical procedure.

Florescent Imaging Cetuximab is a chimeric (mouse/human) monoclonal antibody that targets the epidermal growth factor (EGF) receptor (EGFR). EGFR is highly-expressed in pancreatic ductal adenocarcinoma (PDAC) and is a good target for antibody-mediated imaging, due to its transmembrane position. Cetuximab-IRDye 800CW is cetuximab labeled with IRDye800, an N-hydroxysuccinimide (NHS) ester infrared dye. IRDye800 has very similar properties compared to indocyanine green, and indocyanine green is readily detectable with a number of imaging systems. This study evaluates the Cetuximab-IRDye 800CW as a intraoperative labeling agent.

Patients receive Cetuximab-IRDye 800CW intravenously (IV) at 50 mg or 100 mg over 30 minutes to 1 hour on day 0. Within 2 to 5 days, patients undergo surgery with intraoperative imaging. Cetuximab-IRDye 800CW is used as part of a tumor-targeted molecular imaging procedure operating on the principles of differential accumulation of the antibody-dye conjugate in pancreatic tumor tissue vs normal pancreatic tissue vs pancreatitis tissue.

Excised tissues are prepared as formalin-fixed paraffin-embedded (FFPE) blocks for assessment of fluorescent intensity.

Photoacoustic imaging (PAI) For purposes of non-quantitative comparison, photoacoustic imaging (PAI) of the tumor lesions is also conducted. PAI refers to a non-invasive evaluation by ultrasound of the area of the resected tumor and surrounding tissue. PAI may have special utility for detecting tumors within 5 to 7 mm of depth, with a high degree of spatial resolution, which might be useful to enhance generation of tumor-free surgical margins. PAI does not utilize ionizing radiation, and should complement and conform to the findings from the fluorescent imaging.

PRIMARY OBJECTIVE:

Determine the efficacy of cetuximab-IRDye800 in intraoperatively identifying pancreatic cancer compared to surrounding normal pancreatic and extrapancreatic tissue, as measured by tumor-to-background ratio.

SECONDARY OBJECTIVE:

Determine the tolerability of the cetuximab IRDye800 as an imaging agent in patients undergoing resection of pancreatic cancer.

ELIGIBILITY:
INCLUSION CRITERIA

* Clinically suspected or biopsy confirmed diagnosis of pancreatic adenocarcinoma
* Planned standard of care surgery with curative intent for pancreatic adenocarcinoma
* ≥ 19 years of age
* Life expectancy of more than 12 weeks
* EITHER

  * Karnofsky performance status of at least 70%, OR
  * Eastern Cooperative Oncology Group (ECOG)/Zubrod level 1
* Hemoglobin ≥ 9 gm/dL
* Platelet count ≥ 100,000/mm^3
* Magnesium > the lower limit of normal (LLN) per institution normal lab values
* Potassium > LLN
* Calcium > LLN
* Thyroid-stimulating hormone (TSH) < 13 micro International units/mL

EXCLUSION CRITERIA

* Received an investigational drug within 30 days prior to first dose of cetuximab IRDye800
* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); or unstable angina within 6 months prior to enrollment
* History of infusion reactions to cetuximab or other monoclonal antibody therapies
* Pregnant or breastfeeding
* Evidence of QT prolongation on pretreatment electrocardiography (ECG) (greater than 440 ms in males or greater than 450 ms in females)
* Lab values that in the opinion of the primary surgeon would prevent surgical resection
* Patients receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04-24 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Poultsides, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenthal EL, Kulbersh BD, King T, Chaudhuri TR, Zinn KR. Use of fluorescent labeled anti-epidermal growth factor receptor antibody to image head and neck squamous cell carcinoma xenografts. Mol Cancer Ther. 2007 Apr;6(4):1230-8. doi: 10.1158/1535-7163.MCT-06-0741. PMID 17431103
- [Background] Rosenthal EL, Kulbersh BD, Duncan RD, Zhang W, Magnuson JS, Carroll WR, Zinn K. In vivo detection of head and neck cancer orthotopic xenografts by immunofluorescence. Laryngoscope. 2006 Sep;116(9):1636-41. doi: 10.1097/01.mlg.0000232513.19873.da. PMID 16954995
- [Result] Tummers WS, Miller SE, Teraphongphom NT, Gomez A, Steinberg I, Huland DM, Hong S, Kothapalli SR, Hasan A, Ertsey R, Bonsing BA, Vahrmeijer AL, Swijnenburg RJ, Longacre TA, Fisher GA, Gambhir SS, Poultsides GA, Rosenthal EL. Intraoperative Pancreatic Cancer Detection using Tumor-Specific Multimodality Molecular Imaging. Ann Surg Oncol. 2018 Jul;25(7):1880-1888. doi: 10.1245/s10434-018-6453-2. Epub 2018 Apr 17. PMID 29667116
- [Derived] Lwin TM, Hoffman RM, Bouvet M. The future of tumour-specific fluorescence-guided surgery for pancreatic cancer. Lancet Gastroenterol Hepatol. 2020 Aug;5(8):715-717. doi: 10.1016/S2468-1253(20)30123-0. Epub 2020 May 14. No abstract available. PMID 32416765

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab IRDye800, 50 mg | Cetuximab IRDye800, 100 mg
Started | 6 | 2
Completed | 5 | 2
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab IRDye800, 50 mg | Cetuximab IRDye800, 100 mg | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (7.9) | 70.4 (7.1) | 65.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Peri-operative Cetuximab-IRDye800 Fluorescent Imaging, Both Doses
Description: Cetuximab-IRDye800 (50 mg or 100 mg) was administered pre-operatively, and the uptake of the dye was assessed by observed fluorescence intra-operatively (ie, in vivo) and post-operatively (ex vivo, or "back table"), in tumorous (tumor or tumor-bearing lymph nodes) or normal (non-tumorous) tissues. Collectively, intra-operative and immediately post-operative are considered "peri-operative." The outcome tumor-to-background ratio (TBR) is measured as the mean of the ratios observed between tumor and normal tissue for the participants, and the outcome is expressed as the mean with standard deviation.
Time Frame: up to 5 days
Population: Due to small numbers and the expression of the outcome value as a mean of ratios, the analysis was conducted on all evaluable participants as a single cohort in order to reduce variance/dispersion.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Cetuximab IRDye800, 50 mg: On day 0, participants receive a 100 mg cetuximab loading dose by intravenous infusion (IV), followed 1 hour later by cetuximab-IRDye 800CW IV at 50 or 100 mg, followed by surgery with intraoperative imaging within 2 to 5 days.
  Cetuximab-IRDye800: Administered intravenously (IV) at 50 or 100 mg
  Cetuximab: Administered as a 100 mg IV loading dose
Arm/Group | Cetuximab IRDye800, 50 mg
Number analyzed (Participants) | 6
ratio
  In vivo (tumor at resection): number analyzed (Participants) | 4
  In vivo (tumor at resection) | 2.3 (0.72)
  In vivo (lymph node at resection): number analyzed (Participants) | 2
  In vivo (lymph node at resection) | 6.3 (0.82)
  Ex vivo (post-operative, back-table) | 3.4 (0.4)

2. Secondary Outcome: Cetuximab-IRDye800 Labeling Intensity in Tumor and Non-Tumor Tissues (Ex Vivo)
Description: Cetuximab-IRDye800 (50 mg or 100 mg) florescence intensity was assessed in normal pancreatic tissue; pancreatitis tissue; and pancreatic tumor tissue prepared as formalin-fixed paraffin-embedded (FFPE) blocks. Fluorescent intensity was measured in the image for each tissue, and expressed as counts per pixel. The outcome is expressed for each tissue as the dose-independent mean counts/pixel for the cohort. The outcome is expressed as the mean counts/pixel with standard deviation.
Time Frame: up to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: counts per pixel
Arm/Group | Cetuximab IRDye800, 50 mg
Number analyzed (Participants) | 6
counts per pixel
  Normal pancreatic tissue | 0.02 (0.01)
  Pancreatitis tissue | 0.04 (0.02)
  Pancreatic tumor tissue | 0.09 (0.06)

3. Secondary Outcome: Effect of Cetuximab-IRDye800 Dose on Fluorescence Intensity
Description: Cetuximab-IRDye800 (50 mg or 100 mg) florescence intensity was assessed in normal pancreatic tissue; pancreatitis tissue; and pancreatic tumor tissue prepared as formalin-fixed paraffin-embedded (FFPE) blocks. Fluorescent intensity was measured in the image for each tissue, and expressed as counts per pixel. The outcome is expressed for each tissue as the dose-independent mean fluorescent intensity (MFI) for the cohort. The outcome is expressed as a mean with standard deviation, by dose.
Time Frame: up to 14 days
Population: Tissue sampling and labeling can be imprecise, and there may not have been residual tissue after standard-of-care pathological analysis. Data were not obtained for all participants.
Measure: Mean (Standard Deviation); unit: counts per pixel
Groups:
- Cetuximab IRDye800, 50 mg: On day 0, participants receive a 100 mg cetuximab loading dose by intravenous infusion (IV), followed 1 hour later by cetuximab-IRDye 800CW IV at 50 mg, followed by surgery with intraoperative imaging within 2 to 5 days.
  Cetuximab-IRDye800: Administered intravenously (IV) at 50 mg
  Cetuximab: Administered as a 100 mg IV loading dose
- Cetuximab IRDye800, 100 mg: On day 0, participants receive a 100 mg cetuximab loading dose by intravenous infusion (IV), followed 1 hour later by cetuximab-IRDye 800CW IV at 100 mg, followed by surgery with intraoperative imaging within 2 to 5 days.
  Cetuximab-IRDye800: Administered intravenously (IV) at 100 mg
  Cetuximab: Administered as a 100 mg IV loading dose
Arm/Group | Cetuximab IRDye800, 50 mg | Cetuximab IRDye800, 100 mg
Number analyzed (Participants) | 4 | 2
counts per pixel
  Normal pancreatic tissue | 0.02 (0.01) | 0.03 (0.02)
  Pancreatitis tissue | 0.03 (0.02) | 0.06 (0.03)
  Pancreatic tumor tissue | 0.09 (0.06) | 0.10 (0.05)

4. Secondary Outcome: Sensitivity and Specificity of Ex Vivo Fluorescent Imaging
Description: Sensitivity is the ability of a test to correctly identify patients with the condition, ie, how well Cetuximab-IRDye800 fluorescent imaging detects true-positive patients. Sensitivity is defined as [TP/(TP+FN)], where TP=true-positive, and FN=false-negative. The outcome is a % without dispersion. A higher % means a greater probability that an imaging target identified as cancerous is confirmed by histology to be cancerous, and a lower % means reduced confidence in that result.
  Specificity is the ability of a test to correctly identify patients who do not have the condition, ie, how well Cetuximab-IRDye800 fluorescent imaging detects true-negative patients. Specificity is defined as [TN/(TN+FP)], where TN=true-negative, and FP=false-positive. The outcome is a % without dispersion. A higher % means a greater probability that an imaging target identified as non-cancerous is confirmed by histology to be non-cancerous, and a lower % means reduced confidence in that result.
Time Frame: up to 14 days
Population: Outcome results for sensitivity and specificity of fluorescent imaging were available by dose, and compiled across both doses. Tissue sampling and labeling can be imprecise, and there may not have been residual tissue after standard-of-care pathological analysis. Data were not obtained for all participants.
Measure: Number; unit: percentage of lymph nodes
Units Other Than Participants: Lymph nodes
Groups:
- Cetuximab IRDye800, Both Doses: On day 0, participants receive a 100 mg cetuximab loading dose by intravenous infusion (IV), followed 1 hour later by cetuximab-IRDye 800CW IV at 100 mg, followed by surgery with intraoperative imaging within 2 to 5 days.
  Cetuximab-IRDye800: Administered intravenously (IV) at 50 or at 100 mg
  Cetuximab: Administered as a 100 mg IV loading dose
Arm/Group | Cetuximab IRDye800, 50 mg | Cetuximab IRDye800, 100 mg | Cetuximab IRDye800, Both Doses
Number analyzed (Participants) | 4 | 2 | 6
Number analyzed (Lymph nodes) | 72 | 72 | 144
percentage of lymph nodes
  Sensitivity | 100.0 | 88.2 | 96.1
  Specificity | 78.0 | 32.1 | 67.0

5. Secondary Outcome: Cetuximab-IRDye800 Tumor Detection in Lymph Nodes
Description: Cetuximab-IRDye800 (50 mg or 100 mg) florescence intensity was assessed in excised lymph nodes (ie, ex vivo) that were histologically-determined to be normal or tumor-bearing. Fluorescent intensity was measured in the image for each lymph using close-field fluorescence imaging and expressed as counts per pixel. The outcome is expressed for each tissue as the dose-independent mean fluorescent intensity (MFI) for the cohort. The outcome is expressed as the mean MFI with standard deviation.
Time Frame: up to 14 days
Population: The relationship of the number of participants to number of analyzed lymph nodes (tumor-bearing or not) is not 1:1, & tissue sampling & labeling are imprecise. Participants could contribute none or multiple normal and tumor-bearing lymph node for analysis. Data were not obtained for all participants.
Measure: Mean (Standard Error); unit: counts per pixel
Units Other Than Participants: Lymph nodes
Arm/Group | Cetuximab IRDye800, 50 mg | Cetuximab IRDye800, 100 mg
Number analyzed (Participants) | 4 | 2
Number analyzed (Lymph nodes) | 72 | 72
counts per pixel
  Tumor-bearing lymph nodes: number analyzed (Lymph nodes) | 8 | 16
  Tumor-bearing lymph nodes | 0.071 (0.01) | 0.046 (0.007)
  Histologically normal lymph nodes: number analyzed (Lymph nodes) | 64 | 56
  Histologically normal lymph nodes | 0.018 (0.001) | 0.035 (0.004)

6. Secondary Outcome: Signal-to-Noise Ratio (SNR) by Ex Vivo Photoacoustic Imaging (PAI)
Description: Photoacoustics were assessed as the signal-to-noise ratio (SNR), a unit-less number, as observed for tumor vs surrounding tissue using an ultrasound device. The value observed for tumor tissue is considered signal, and the value for normal tissue is considered noise. The more the ratio is greater than 1 reflects the more that the tumor tissue reflects an ultrasound signal compared to normal tissue. The outcome is expressed as the ratio of mean SNR signal for tumor tissue to normal tissue, without dispersion.
Time Frame: up to 5 days
Population: Tissue sampling and labeling can be imprecise. Due to small numbers and the expression of the outcome value as a mean of ratios, the analysis was conducted on all evaluable participants as a single cohort. Data were not obtained for all participants. Dispersion was not and can not be determined for the outcome, a ratio (ratio of means).
Measure: Number; unit: ratio
Arm/Group | Cetuximab IRDye800, 50 mg
Number analyzed (Participants) | 4
ratio | 3.7

7. Secondary Outcome: Signal-to-Noise Ratio (SNR) by In Vivo Photoacoustic Imaging (PAI)
Description: Photoacoustic imaging (PAI) was to be used to evaluate tumor and normal margin tissues (waste tissue) immediately peri-operatively (in vivo) and prior to pathological evaluation. The signal-to-noise ratio (SNR) as measured in dB of the tumor was to be calculated in the tumor specimens for comparison to surrounding normal tissue. The outcome would be expressed as the mean of the ratios, with standard deviation, and data used to qualitatively confirm the findings with Cetuximab-IRDye 800CW fluorescent imaging.
Time Frame: up to 5 days
Population: The in vivo photoacoustic imaging (PAI) component of this study was not IRB-approved, and this part of the study was not conducted.
Arm/Group | Cetuximab IRDye800, 50 mg | Cetuximab IRDye800, 100 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Toxicity (≥ Grade 2)
Description: Toxicity was assessed as the number of grade 2 or greater adverse events [Common Terminology Criteria for Adverse Events (CTCAE) version 4.03] determined to be clinically-significant and definitely-, probably-, or possibly-related to cetuximab-IRDye 800CW.
  The outcome is reported as the number of treatment-related adverse events ≥ grade 2 without dispersion, by dose level.
Time Frame: Up to 30 days
Measure: Number; unit: Adverse events
Arm/Group | Cetuximab IRDye800, 50 mg | Cetuximab IRDye800, 100 mg
Number analyzed (Participants) | 6 | 2
Adverse events | 1 | 0

ADVERSE EVENTS:
Time Frame: 30 days +- one week
Arm/Group | Cetuximab IRDye800, 50 mg | Cetuximab IRDye800, 100 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab IRDye800, 50 mg (N=6) | Cetuximab IRDye800, 100 mg (N=2)
Pancreatic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab IRDye800, 50 mg (N=6) | Cetuximab IRDye800, 100 mg (N=2)
Anemia (Blood and lymphatic system disorders) | 5 (16) | 2 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (10) | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (12) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 0 (0)
Weight loss (Investigations) | 2 (3) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (10) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (19) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (19) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (9) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (10) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 4 (9) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT02736578/Prot_SAP_000.pdf